CLINICAL TRIAL: NCT00255788
Title: A Randomized Phase II Study of Two Different Schedules of RAD001C in Patients With Recurrent/Metastatic Breast Cancer
Brief Title: Everolimus in Treating Patients WIth Recurrent or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I163; CAN-NCIC-IND163 (Other: PDQ); NOVARTIS-CAN-NCIC-IND163 (Other: Novartis); CDR0000450849 (Other: PDQ)
Record Dates: First submitted 2005-11-18; First posted 2005-11-21 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IV breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator): Everolimus - 28 days q 4 wk
  Interventions: Drug: everolimus
- Arm B (Active Comparator): Everolimus - days 1, 8, 15 and 22 q 4wks
  Interventions: Drug: everolimus

INTERVENTIONS:
Drug: everolimus

SUMMARY:
RATIONALE: Everolimus may stop the growth of tumor cells by blocking blood flow to the tumor.

PURPOSE: This randomized phase II trial is studying two different schedules of everolimus to see how well they work in treating patients with recurrent or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of 2 different treatment schedules of everolimus, in terms of clinical/radiological response and early progression, in patients with recurrent or metastatic breast cancer.

Secondary

* Determine the time to progression and response duration in patients treated with these regimens.
* Determine the toxic effects of these regimens in these patients.
* Correlate molecular markers of mTOR activity in tumor tissue with objective tumor response in patients treated with these regimens.

OUTLINE: This is a randomized, open label, multicenter study. Patients are stratified according to presence of visceral metastases (yes vs no) and prior chemotherapy regimens for recurrent disease (0 vs 1). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral everolimus once daily on days 1-28.
* Arm II: Patients receive oral everolimus on days 1, 8, 15, and 22. In both arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 4 weeks and then periodically until disease progression.

PROJECTED ACCRUAL: A total of 60 patients (30 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Metastatic or recurrent disease
  * Considered incurable
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral CT scan
* Two primary breast cancers allowed
* Paraffin-embedded primary or metastatic tumor sample available
* No known brain metastases
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Sex

* Male or female

Menopausal status

* Not specified

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN

Renal

* Creatinine ≤ 1.5 times ULN

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active uncontrolled infection
* No upper gastrointestinal condition or other condition that would preclude ability to take oral medication
* No other serious medical condition that would preclude study participation
* No psychiatric illness or neurologic disorder that would preclude study compliance
* No other malignancy within the past 5 years except curatively treated nonmelanoma skin cancer or carcinoma in situ of the cervix or bladder

PRIOR CONCURRENT THERAPY:

Chemotherapy

* At least 4 weeks since prior chemotherapy
* Prior adjuvant chemotherapy allowed
* No more than 1 prior chemotherapy regimen for metastatic or recurrent disease

Endocrine therapy

* At least 5 days since prior hormonal therapy

Radiotherapy

* At least 4 weeks since prior radiotherapy except for low-dose, limited-fraction, palliative, nonmyelosuppressive radiotherapy, defined as radiotherapy to < 20% of functioning bone marrow
* If prior radiotherapy was to sole site of disease, must have subsequent documented disease progression at that site

Surgery

* At least 3 weeks since prior major surgery

Other

* Concurrent prophylactic bisphosphonates allowed, if started prior to study entry
* No concurrent potent inhibitors of cytochrome 3A4, such as erythromycin, diltiazem, or ketoconazole and similar antifungals
* No other concurrent anticancer therapy
* No other concurrent investigational agents
* No concurrent grapefruit juice

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2005-05-10 (Actual); Primary Completion 2008-07-22 (Actual); Study Completion 2011-01-18 (Actual)

PRIMARY OUTCOMES:
Response rate by clinical evaluation every 4 weeks and radiologic reevaluation every 8 weeks
Early progression rate by clinical evaluation every 4 weeks and radiologic reevaluation every 8 weeks

SECONDARY OUTCOMES:
Adverse event rates
Time to progression by clinical evaluation every 4 weeks and radiologic reevaluation every 8 weeks
Response duration by evaluation 4 weeks after response and then every 8 weeks
Correlative assessment of response with molecular markers of mTor activity on archival tissue
Optional correlative assessment of response with molecular markers of mTor activity on fresh tissue

CONTACTS AND LOCATIONS:
Overall Officials: Susan Ellard, MD, Study Chair — British Columbia Cancer Agency - Centre for the Southern Interior; Karen A. Gelmon, MD, Study Chair — British Columbia Cancer Agency
Locations (5):
- Canada (5):
  - British Columbia Cancer Agency - Centre for the Southern Interior, Kelowna, British Columbia
  - Fraser Valley Cancer Centre at British Columbia Cancer Agency, Surrey, British Columbia
  - British Columbia Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Toronto Sunnybrook Regional Cancer Centre at Sunnybrook and Women's College Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ellard SL, Clemons M, Gelmon KA, Norris B, Kennecke H, Chia S, Pritchard K, Eisen A, Vandenberg T, Taylor M, Sauerbrei E, Mishaeli M, Huntsman D, Walsh W, Olivo M, McIntosh L, Seymour L. Randomized phase II study comparing two schedules of everolimus in patients with recurrent/metastatic breast cancer: NCIC Clinical Trials Group IND.163. J Clin Oncol. 2009 Sep 20;27(27):4536-41. doi: 10.1200/JCO.2008.21.3033. Epub 2009 Aug 17. PMID 19687332